CLINICAL TRIAL: NCT02604108
Title: Training Program for Happy Family Kitchen Movement, A Community-based Research to Enhance Family Health, Happiness and Harmony in Hong Kong
Brief Title: Training Program for Happy Family Kitchen Movement Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Council of Social Service (Other); The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Project Manager (Health Communication), The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW15-083
Record Dates: First submitted 2015-11-05; First posted 2015-11-13 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Physical Activity; Healthy Diet; Family Health, Happiness and Harmony; Quality of Life
Keywords: physical activity; healthy diet
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Exercise (Experimental): Physical Exercise: Participants will receive training and health messages on positive psychology and healthy living style focusing on physical activity.
  Interventions: Behavioral: Physical Exercise
- Healthy Diet (Experimental): Healthy Diet: Participants will receive training and health messages on positive psychology and healthy living style focusing on healthy diet.
  Interventions: Behavioral: Healthy Diet

INTERVENTIONS:
Behavioral: Physical Exercise — The Physical Exercise arm includes a training workshop and electronic health messages related to positive psychology and physical activity for all participants in physical exercise group. Skills on program design and implementation will be conducted for those participants, who will design and implement community-based family intervention to the public.
  The training workshop includes: (i) 2-day core session and half day booster session for trainers; and (ii) 1-day core session and half day booster session for ambassadors
  Arms: Physical Exercise
Behavioral: Healthy Diet — The Healthy Diet arm includes a training workshop and electronic health messages related to positive psychology and health diet for all participants in healthy diet group. Skills on program design and implementation will be conducted for those participants, who will design and implement community-based family intervention to the public.
  The training workshop includes: (i) 2-day core session and half day booster session for trainers; and (ii) 1-day core session and half day booster session for ambassadors
  Arms: Healthy Diet

SUMMARY:
This training program is a part of Happy Family Kitchen Movement Project, which is a community-based research project with 3 main components for data collection - training programs, community-based family interventions and public education events. The training program involves various organizations, including non-government organizations and schools across districts in different regions of Hong Kong.

In the study, the investigators would use training programs as a capacity building method and an essential media delivering the holistic health knowledge (positive psychology, physical activity, healthy diet) to the public. The project team will provide training program for the participants, including: (i) train-the-trainer workshops for the social service workers, who will conduct community-based family intervention programs; and (ii) train-the-trainer ambassadors for the volunteers who may assist to implement health-related activities for the public.

DETAILED DESCRIPTION:
In recent years, Hong Kong is undergoing rapid changes together with macro social and economic trends. Demographic shifts, both immigration across national borders and migration with nations, as well as the changing in societal norms and values have significant impact on the structures and relationships within families. Physical inactivity was found to be a local and worldwide issue and most Hong Kong people are having a sedentary lifestyle . Studies show that the increase of physical activity and healthy diet reduce the risk of chronic diseases, and improve cardio-pulmonary functions; whereas sedentary behaviors increase the risk. Positive psychology is used as a preventive and complementary medicine, which also is crucial component in family holistic health (happiness, harmony and health). Positive psychology aims to focus on positive emotions, and uses scientific understanding to implement effective intervention, which lead to positive attitudes, happiness and fulfillment. Positive psychology interventions can be effective in the enhancement of subjective and psychological well-being and may help to reduce depressive symptom levels.

The increasingly complex and diverse family structure is leading to a major concern in the well-being of families in Hong Kong, including their health, happiness and harmony (3Hs). Family life and health education should be strengthened to meet the increasing needs of healthy lifestyle among Hong Kong families. A framework of "Five principles of positive psychology" to enhance family communication was developed in Family Kitchen I project, which is the sub-project of FAMILY Project. The five principles concerned are happiness, flow, gratitude, savoring, and health. It used "eating" and "kitchen" as a platform to develop a positive environment for family well-being and communication, which based on five positive psychology approaches to improve communication in the family, and in turn promote FAMILY Health, Happiness and Harmony (3Hs).

Following the theme on FAMILY 3Hs, the new work focus is to promote family holistic health with emphasize on the interaction and integration of physical and psychosocial health. In light of these concerns, FAMILY projects - Happy Family Kitchen Movement (HKFM) project will be conducted at territory-wide level. HKFM project is to focus on "FAMILY Holistic Health" and aims at promoting higher level of physical activity and healthy diet for people of all ages. It also enhances family interaction, pleasure and well-being, as well as FAMILY 3Hs. HKFM is a community-based research project with 3 main components - training program, community-based family intervention and public education event.

Train-the-trainer workshop would be provided to the service workers and ambassadors in different districts to equip them with knowledge and skills in implementing the community-based family intervention programs.

In the current study, the investigators would use training workshops as a capacity building method and an essential media delivering the knowledge on holistic health.to the public. The holistic health information is related to positive psychology, physical activity and healthy diet.

The project team will provide training workshops for the participants, including: (i) train-the-trainer workshops for the social service workers, who will conduct community-based family intervention programs; and (ii) train-the-ambassador workshops for the ambassadors who will assist the social service workers to implement health-related activities for the public.

Need assessment and focus group interview will be conducted before program design and after conducting the training, respectively. Process evaluation will be performed to evaluate the process of each component of the program. Qualitative and quantitative evaluations will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Chinese speaking;
* Able to complete study questionnaire;
* Aged 18 or above.

Exclusion Criteria:

* Do not fit the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in knowledge in relation to positive psychology, physical activity, and healthy diet | Baseline, 6 weeks
  Change in knowledge in relation to positive psychology, physical activity, and healthy diet will be assessed by outcome-based questionnaire

SECONDARY OUTCOMES:
Change in knowledge in relation to positive psychology, physical activity, and healthy diet | Baseline, immediately after core session , 6 weeks, 3 months
  Change in knowledge in relation to positive psychology, physical activity, and healthy diet will be assessed by outcome-based questionnaire
Change in attitude on incorporating positive psychology, physical activity, and healthy diet in community-based interventions | Baseline, immediately after core session, 6 weeks, 3 months
  Change in attitude on incorporating positive psychology, physical activity, and healthy diet in community-based interventions will be assessed by outcome-based questionnaire
Change in attitude on practicing positive psychology, physical activity, and healthy diet | Baseline, immediately after core session, 6 weeks, 3 months
  Change in attitude on practicing positive psychology, physical activity, and healthy diet will be assessed by outcome-based questionnaire
Change in personal holistic health behavior in relation to positive psychology, physical activity, and healthy diet | Baseline, 2 weeks, 6 weeks, 3 months
  Change in personal holistic health behavior in relation to positive psychology, physical activity, and healthy diet will be assessed by behavior indicator scales
Change in family holistic health behavior in relation to positive psychology, physical activity, and healthy diet | Baseline, 2 weeks, 6 weeks, 3 months
  To compare the family holistic health behavior in relation to positive psychology, physical Change in family holistic health behavior in relation to positive psychology, physical activity, and healthy diet will be assessed by behavior indicator scales
Change in knowledge sharing with family members in relation to positive psychology, physical activity, and healthy diet | Baseline, 2 weeks, 6 weeks, 3 months
  Change in knowledge sharing with family members in relation to positive psychology, physical activity, and healthy diet will be assessed by outcome-based questionnaire
Change in personal happiness | Baseline, 6 weeks, 3 months
  Subjective happiness will be assessed by subjective happiness scale
Changes in personal health | Baseline, 6 weeks, 3 months
  Personal health will be assessed by outcome-based questionnaire
Changes in quality of life | Baseline, 6 weeks, 3 months
  The quality of life will be assessed by SF-12 v2 health survey
Changes in family health, happiness, and harmony (3Hs) | Baseline, 6 weeks, 3 months
  Family 3Hs will be assessed by the family well-being scale
Changes in physical fitness [grip strength (kg), chair stand (times), single leg stand (s), seat and reach (cm)] | Baseline, 6 weeks
  Physical fitness will be assessed by simple physical tests
Satisfaction toward training program | immediately after core session, immediately after 6-week booster session
  Satisfaction towards training session will be assessed by a program evaluation measure
Changes in body fat and body weight | Baseline, 6 weeks
  Changes in body fat and body weight will be assessed by a standard body fat measuring scale

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, DN, Principal Investigator — The University of Hong Kong; Tai Hing Lam, MD, Study Chair — The University of Hong Kong; Henry CY Ho, PhD, Study Director — The University of Hong Kong
Locations (1):
- The Hong Kong Council of Social Service, Wan Chai, Hong Kong, China

REFERENCES:
- [Background] Yoshikawa H. Integrating methods in the science of family health: new directions from an institute of medicine workshop report. Arch Pediatr Adolesc Med. 2012 Jul 1;166(7):659-61. doi: 10.1001/archpediatrics.2012.510. No abstract available. PMID 22751883
- [Background] Hu FB. Globalization of diabetes: the role of diet, lifestyle, and genes. Diabetes Care. 2011 Jun;34(6):1249-57. doi: 10.2337/dc11-0442. PMID 21617109
- [Background] Seligman ME, Csikszentmihalyi M. Positive psychology. An introduction. Am Psychol. 2000 Jan;55(1):5-14. doi: 10.1037//0003-066x.55.1.5. PMID 11392865
- [Background] Sin NL, Lyubomirsky S. Enhancing well-being and alleviating depressive symptoms with positive psychology interventions: a practice-friendly meta-analysis. J Clin Psychol. 2009 May;65(5):467-87. doi: 10.1002/jclp.20593. PMID 19301241